CLINICAL TRIAL: NCT03326219
Title: Histopathological Study of the Vena Saphena Magna After Mechanochemical Endoveneous Ablation
Brief Title: Endoveneous Histologic Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty finding eligible patients
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Michel Reijnen, Dr. Michel Reijnen, MD, PI, vascular surgeon, Rijnstate Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL38948.091.12
Record Dates: First submitted 2017-10-13; First posted 2017-10-31 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Varicose Veins
Keywords: MOCA; VSM; Clarivein; Histological
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aethoxysklerol clarivein during leg amp (Other): Clarivein treatment with Aethoxysklerol in 5 patients during lower or upper leg amputation
  Interventions: Procedure: Clarivein

INTERVENTIONS:
Procedure: Clarivein — The Clarivein technique uses mechanical damage to the endothelium of the vein wall through a rotating tip of the catheter. At the same time a sclerosans is injected, causing occlusion of the vein. No heating is used in this technique .

SUMMARY:
A new technique, mechanochemical endovenous ablation (MOCA), using the ClariVein ® system is recently developed. To date, histopathological data after mechanochemical endovenous ablation are not known.

The aim of this study is the histopathological analysis of venous injury using mechanochemical endovenous ablation.

DETAILED DESCRIPTION:
Background:

Varicose veins are a common problem in the Western world. Epidemiological studies show that one quarter of adults have some form of varicose veins. Women are two to three times more affected than men. The prevalence of varicose veins increases steadily with age and is among the top ten of the complaints that people visit their General Practitioner. The main risk factors are prolonged standing or sitting, pregnancy, gender and age. The symptoms of varicose veins are variable and range from cosmetic complaints to venous ulcers.

Stripping of the great saphenous vein(GSV) has been the golden standard for GSV insufficiency for a long time. It is performed under regional or general anesthesia and has a high recurrence rate of 18-40% at 5 years. In addition, the procedure leads to significant postoperative symptoms, especially pain, hematoma and the risk of injury to the saphenous nerve.

In recent years, endovenous techniques have been developed for the treatment of primary GSV insufficiency. Particularly laser endovenous ablation (EVLA) and radiofrequency ablation (VNUS) became accepted technologies and are widely applied in practice. These thermal-based techniques have the advantage that the surgery can be performed with local anesthesia. In addition, endovenous techniques cause less hematoma, pain, and have superior cosmetics and earlier resumption of normal activities/work compared to the conventional surgical stripping.

Endothermal techniques use heat, which has potential risk to damage surrounding tissues. For this reason, patients are treated with tumiscence anesthesia, requiring multiple punctures around the vein. Most patients experience tumiscence anesthesia as unpleasant. Despite the tumiscence anesthesia, patients may still observe postoperative pain, which may last for weeks.

Laser energy is absorbed and converted into intraluminal heat. This process causes steam bubbles, as described by Proebstle. In previous studies, intraluminal and extraluminal temperature measurements were done during endovenous laser ablation. In addition, acute pathological changes after endovenous laser ablation is studied in a recent study. The loss of laser energy was confined to the inner part of the media. No perivascular damage was seen. However, 1% of patients treated with endovenous laser ablation has nerve damage or paresthesias. It suggests that perivascular damage to some extent still exists.

The effects of foam sclerosis appear to be limited to the endothelium and tunica media of the vein wall. Pathological changes occur rapidly within the first 2 minutes after treatment. After 30 minutes intimal detachment of the tunica media, and the formation of microthrombi are detected. The addition of a balloon injury of the vessel wall prior to foam sclerosis, results in a higher percentage of endothelial damage. However, in practice, the clinical results of foam sclerosis disappointing. The occlusionrate from 1 to 5 years were 81 and 73% in a recent meta-analysis.

A new technique, mechanochemical endovenous ablation (MOCA), using the ClariVein ® system is recently developed. The first studies show that MOCA a safe and effective treatment for varicose veins. This technique uses mechanical damage to the endothelium of the vein wall through a rotating tip of the catheter. At the same time a sclerosans is injected, causing occlusion of the vein. No heating is used in this technique . Tumiscence anesthesia is redundant and complications that occur in thermal endovenous techniques, such as pain, hematoma formation, induration and paresthesias could be reduced. To date, histopathological data after mechanochemical endovenous ablation are not known.

Objective of the study:

The aim of this study is the histopathological analysis of venous injury using mechanochemical endovenous ablation

Study design:

The Endovenous Histology study is a histopathological study on the effects of mechanochemical endovenous ablation. The studycentre will be:

- Rijnstate Hospital, Arnhem.

5 patients with irreversible tissue damage to the lower extremities based on atherosclerotic peripheral vascular disease will be included in the study Endovenous Histology, after signing informed consent. All patients included, are scheduled for an elective upper or underleg amputation. The preprocedural status will be determined by height, weight, comorbidities, ASA classification, medications, previous vascular surgery and venous duplex of the VSM.

Subsequently 5 patients are treated with MOCA of the VSM to the amputation level prior to the amputation under general or spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Elective indication for leg amputation
2. Peripheral arterial disease
3. Age > 18 years
4. Written informed consent

Exclusion Criteria:

1. Patient is incapable of informed consent
2. Pregancy and lactation
3. Previous surgical or endovenous treatment of the greater saphenous vein in the amputed leg
4. Great saphenous vein is used for bypass surgery
5. INR > 1.8
6. ASA 5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Occlusion of the with Clarivein treated vein | 2 years of inclusion and analyzation
  Occlusion of the with the Clarivein (Aethoxysklerol) treated vein, check wheter or not treatment was succesfull.
Depth of damage inside and/or outside the venous wall | 2 years of inclusion and analyzation
  Depth of damage inside and/or outside the venous wall is to check whether or not the venous wall is damaged due to the Clarivein treatment

SECONDARY OUTCOMES:
Analysis of intraluminal clot / scar | 2 years of inclusion and analyzation
  After excision of the treated vein of the amputated leg it will be analysed on intraluminal clot/scar
Morphological changes of the saphenous nerve due to damage of treatment | 2 years of inclusion and analyzation
  Analyses of the changes of the saphenous nerve in the treated area (amputated lef) due to the Clarivein treatment.
Perivascular damage resulting from treatment | 2 years of inclusion and analyzation
  Analyses of the perivascular damage in the amputated leg as a result of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: MMPJ Reijnen, MD, Principal Investigator — Rijnstate
Locations (1):
- Rijnstate, Arnhem, Gelderland, Netherlands